CLINICAL TRIAL: NCT01523522
Title: Etude de l'efficacité et de la sécurité d'Injections Intra-sphinctériennes de Myoblastes Autologues Chez Des Patients Atteints d'Incontinence Anale sévère Par Insuffisance sphinctérienne
Brief Title: Autologous Myoblast Intrasphincteric Injection for Fecal Incontinence
Acronym: MIAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/067/HP
Record Dates: First submitted 2012-01-23; First posted 2012-02-01 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Myoblast; Surgery
MeSH Terms: conditions — Fecal Incontinence | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- myoblast injection (Active Comparator): autologous myoblast
  Interventions: Other: Myoblast injection
- saline solution injection (Placebo Comparator): saline solution injection in anal sphincter
  Interventions: Procedure: saline solution injection

INTERVENTIONS:
Other: Myoblast injection — Autologous myoblast injection in the anal sphincter
  Arms: myoblast injection
Procedure: saline solution injection — saline solution injection in anal sphincter
  Arms: saline solution injection

SUMMARY:
This project aims to offer autologous muscle-derived progenitor cell injection as an efficient mini-invasive surgical therapy that would be simple for the patient and could be used in a majority of cases, including in young women in the post-partum. This approach may provide efficient tissue repair of the striated anal sphincter which is not permitted by existing therapies. This innovative therapy may ultimately be proposed after failure of the common treatments and before an high-risk invasive surgical intervention. Besides, injection of muscle-derived progenitor cells in animals has shown very encouraging results of the sphincter function assessed ex vivo. Hence, a high benefit may be expected with this approach.

DETAILED DESCRIPTION:
after verification of information and inclusion criteria. patients were randomized to treatment or placebo arms and receive the injections.

an evaluation of the function and quality of life are realized. after a period of 6 months, patients in the placebo arm receive the injection of myoblasts that have been preserved.

ELIGIBILITY:
Inclusion criteria

* age between 20 and 65 years
* severe fecal incontinence from at least three months
* Jorge et Wexner score ≥ 10
* incontinence refractory to medical treatment and to reeducation from at least three months
* incontinence due to lesion of the external anal sphincter
* incontinence without significant anal sphincter rupture or rupture ≤ 30% of circumference assessed by endo-anal ultra-sonography
* integrity or not of the internal anal sphincter
* fecal incontinence with normal rectum capacity (maximum tolerable volume ≥ 150 ml assessed by ano-rectal manometry)
* fecal incontinence without associated rectal static disorder on defeco-MRI
* fecal incontinence without bilateral complete neuropathy assessed by electro-physiology

Exclusion criteria

* fecal incontinence with rupture > 30 % of the external anal sphincter
* fecal incontinence with bilateral lesions on the sacral nerves
* Crohn's disease or ulcerative colitis
* unstable type 1 or type 2 diabetes
* myopathy
* peripheral or central neurological diseases
* treatment with laxatives, suppositories or enema
* practice of anal intercourse except if stopped during the study
* treatment with immunosuppressive or cytostatic drugs, CoA HMG reductase inhibitors, morphine derivatives
* treatment of constipation or rectal dyschesia
* pregnancy or breast-feeding,lack of effective contraception during the study (female)
* allergy to antibiotics (cephalexin, metronidazole)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Improvement of anal incontinence score | 6 months

SECONDARY OUTCOMES:
Improvement of quality of life score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BOYER, PhD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Rouen University Hospital, Rouen
  - MICHOT, Rouen

REFERENCES:
- [Derived] Bisson A, Le Corre S, Joly-Helas G, Chambon P, Demoulins L, Jean L, Adriouch S, Drouot L, Giverne C, Roussel F, Jacquot S, Doucet C, Michot F, Lamacz M, Frebourg T, Flaman JM, Boyer O. Chromosomal instability but lack of transformation in human myoblast preparations. Cell Transplant. 2014;23(12):1475-87. doi: 10.3727/096368913X670192. PMID 25565635